CLINICAL TRIAL: NCT07211438
Title: Evaluating the Role of Psilocybin Monitors in Psilocybin Therapy for Treatment Resistant Depression: A Pilot Randomized Clinical Trial
Brief Title: Evaluating the Role of Psilocybin Monitors in Psilocybin Therapy for Treatment Resistant Depression
Acronym: PSI-TNT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ishrat Husain, MBBS, MD (Res.), FRCPsych(U.K.), FRCP(C), Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5203
Record Dates: First submitted 2025-10-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Treatment-Resistant Depression
Keywords: Psilocybin; Psychedelics; Treatment resistant depression; Clinical Trial
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psilocybin + Safety Monitoring (PSM) (Experimental): Psilocybin 25 mg plus PSM
  Interventions: Drug: Psilocybin
- Psilocybin + Psychedelic Assisted Therapy (PAT) (Experimental): 25 mg of psilocybin plus PAT
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 25 mg Psilocybin

SUMMARY:
Psilocybin, the chemical component of "magic mushrooms", has been administered with psychological support in several randomized clinical trials (RCTs) showing large and sustained antidepressant effects.

The purpose of this study is to determine the role of psilocybin monitors on the effects of psilocybin therapy in adults with treatment resistant depression.

DETAILED DESCRIPTION:
Psilocybin, the chemical component of "magic mushrooms", has been administered with psychological support in several randomized clinical trials (RCTs) showing large and sustained antidepressant effects.

The purpose of this study is to determine the role of psilocybin monitors on the effects of psilocybin therapy in adults with treatment resistant depression.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 70 years old;
2. Are outpatients;
3. Must be deemed to have capacity to provide informed consent;
4. Must read, sign and date the informed consent form independently. Proxy consent, including consent from a Legally Authorized Representative (LAR), is not permitted in this study;
5. Stated willingness to comply with all study procedures;
6. Ability to read and communicate in English, such that their literacy and comprehension is sufficient for understanding the consent form and study questionnaires, as evaluated by study staff obtaining consent
7. Primary DSM-5 diagnosis of non-psychotic MDD, single or recurrent, and current Major Depressive Episode (MDE) based on the Mini-International Neuropsychiatric Interview (MINI) for DSM-5 administered at the first screening visit;
8. Participants diagnosed with treatment-resistant depression defined as individuals with a baseline HamD-17 score > 14 and that have not responded to two or more separate trials of antidepressants at an adequate dosage and duration (an antidepressant resistance rating score of three or more is considered an adequate trial) based on the Antidepressant Treatment History Form (ATHF) (Sackeim & Sackeim, 2001); there is no upper limit on the number of treatment failures;
9. Ability to take oral medication;
10. Individuals with an eGFR above 40mL/min/1.73m2 and all blood work on clinical laboratory tests assessed as not clinically significant by study delegate physician at Screening (V1)
11. Individuals who are capable of making their partner pregnant or who are capable of becoming pregnant: use of condoms or highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation;
12. Individuals who are willing to and tapered off current antidepressants, antipsychotics, mood stabilizers, ketamine, esketamine, monoaminergic medicines, and stimulants used for augmentation of antidepressant therapy for a minimum of 2-weeks (or more depending on the medication) prior to Baseline (V2) and for the duration of the study and whose prescribing physician confirms that it is safe for them to do so;
13. Individuals who are willing to and have tapered off current inhibitors of 5'-diphospho-glucuronosyltransferase (UGT)1A9 and 1A10, aldehyde dehydrogenase inhibitors (ALDHs) and alcohol dehydrogenase inhibitors (ADHs) for a minimum of 2-weeks (or more depending on the medication) prior to Baseline (V2) and for the duration of the study and whose physician confirms that it is safe for them to do so;
14. Individuals must have a designated caregiver who is able to bring them home after treatment sessions and stay with them for at least 24 hours after psilocybin has been administered;
15. Individuals who are willing to not receive additional psychotherapy outside of the study throughout the active duration of the study; AND
16. Agreement to adhere to Lifestyle Considerations (section 4.5) throughout study duration.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this clinical trial:

1. Pregnant as assessed by a urine pregnancy test at Screening (V1) and Baseline (V2) or individual's that intend to become pregnant during the study or are breastfeeding;
2. Treatment with another investigational drug or other intervention within 30 days of Screening (V1);
3. Brain stimulation treatment within 6 months of Screening (V1);
4. Use of psychedelics within 6 months of Screening (V1);
5. Have initiated psychotherapy in the preceding 4 weeks prior to Screening (V1);
6. Have a DSM-5 diagnosis of moderate to severe substance use disorder (recreational use of tobacco, alcohol, cannabis and prescribed opioids are permitted) within the preceding 6 months;
7. Have active suicidal ideation with intent and plan, certified by the Mental Health Act (MHA), determined by a study physician;
8. Any DSM-5 lifetime diagnosis of mania or hypomania, a schizophrenia-spectrum disorder, obsessive-compulsive disorder, psychotic disorder (unless substance induced or due to a medical condition), bipolar I or II disorder, paranoid personality disorder, borderline personality disorder, or neurocognitive disorder as determined by medical history and the MINI diagnostic interview;
9. Any first-degree relative with a diagnosis of schizophrenia-spectrum disorder; psychotic disorder (unless substance-induced or due to a medical condition), as determined by the family medical history form and discussions with the participant;
10. Presence of a relative or absolute contraindication to psilocybin, including a drug allergy, recent stroke history (within preceding six months) , uncontrolled hypertension (consistent blood pressure readings above 160/100 mmHg: measured twice with one hour between measurements), low blood pressure (blood pressure reading lower than 90/60mmHg), labile blood pressure (defined as episodes of both high and low blood pressure within a 24-hour period), recent myocardial infarction (within preceding six months), all types of cardiac arrhythmia, severe coronary artery disease (symptomatic with chest pain, angina heart palpitations or shortness of breath), or moderate to severe renal impairment (eGFR of below 40 mL/min ) or hepatic impairment (as a Child-Pugh score of B or C, determined through liver function tests);
11. Presence of baseline prolonged QTc (defined as greater than 450 milliseconds (ms) in men and greater than 460 ms in women) or Torsade de Pointes as measured by the ECG or a history of long QTc syndrome or related risk factors ;
12. Any other clinically significant physical illness including chronic infectious diseases or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of evaluating the role of psilocybin monitors in a clinical trial of psilocybin therapy for treatment resistant depression | 24 months
  Percentage of participants recruited, randomized, and retained

SECONDARY OUTCOMES:
Tolerability and safety of administering psilocybin therapy (25 mg) for treatment resistant depression | 24 months
  Type and number of adverse effects or serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ishrat Husain, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - Toronto Western Hospital (University Health Network), Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No